CLINICAL TRIAL: NCT05807386
Title: WE Are Active and In This toGetHer (WEIGH): a Randomised Controlled Trial to Ascertain the Feasibility of a Home-based Exercise Programme for People Living With Overweight and Obesity
Brief Title: Home-Based Exercise for Adults Living With Overweight and Obesity
Acronym: WEIGH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coventry University (Other)
Responsible Party: Principal Investigator, Sofie Power, Principal Investigator, Coventry University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P149993
Record Dates: First submitted 2023-03-07; First posted 2023-04-11 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Overweight and Obesity
Keywords: home-based exercise
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): Participants will undertake a 12 week, online delivered, home-based exercise programme.
  Interventions: Behavioral: Home-based exercise programme
- Waitlist Control (No Intervention): Participants assigned to the waitlist control will adhere to their usual routine.

INTERVENTIONS:
Behavioral: Home-based exercise programme — A 12 week, online delivered, home-based exercise programme.
  Arms: Exercise Intervention

SUMMARY:
The study aims to implement a 12-week home-based exercise programme utilising an online intervention delivery platform. The focus will be on increasing exercise behaviour within the participant's home setting using aerobic, resistance and flexibility exercises as well as behaviour change techniques. Following the programme, semi-structured interviews will be conducted, to explore participant experiences.

It is hypothesised that the exercise programme will be feasible, accessible and acceptable.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥25kg/m² or BMI ≥30kg/m²
* English speaking
* Able to follow visual and verbal instructions
* Access to the internet and accompanying technology (e.g. laptop or tablet)
* Physically able to undertake aerobic, resistance and flexibility exercise

Exclusion Criteria:

* Unable to provide informed consent
* Receiving invasive medical treatment or planned surgery preceding to, or during, the programme
* Severe mental or physical limitations precluding participation safely in the home environment
* No access to the internet and/or facilitative technology such as a laptop or tablet
* Pregnancy
* Current smoker or vaping.
* Currently or very recently stopped taking weight loss medication (within the last two weeks)
* Recently experienced substantial weight change (defined as 5% within 6-12 months)
* Presence of contraindications to exercise
* Pacemaker and/or other implanted metal device
* At high risk of cardiovascular event

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of the programme through recruitment rate | Calculated at trial end, i.e.12 weeks after inclusion.
  Recruitment rate will be calculated by dividing the number of eligible candidates by the number who consent to participate.
Feasibility and acceptability of the programme through attrition | Calculated at trial end, i.e. 12 weeks after inclusion.
  Attrition rate will be defined and calculated as discontinuation of the intervention without return.
Feasibility and acceptability of the programme through adherence | Calculated at trial end, i.e. 12 weeks after inclusion.
  Adherence will calculated by monitoring the online platform engagement and outputs from post exercise session questionnaires.
Feasibility and acceptability of the programme through intervention engagement | Calculated at trial end, i.e. 12 weeks after inclusion.
  Engagement will be calculated by monitoring participant's activity on the online platform.
Feasibility and acceptability of the programme through completion rate | Calculated at trial end, i.e. 12 weeks after inclusion.
  Completion rate will be calculated by dividing the number of participants who successfully complete the programme, by the number of participants that attempt.
Acceptability and experience of the programme via participant interviews | Evaluated after intervention period, i.e. up to 12 weeks after inclusion offer.
  Interviews will take place between the researcher and participant to explore their experience on the programme and identifying areas for improvement. This may be with participants who completed the intervention, withdrew or declined to participate.

SECONDARY OUTCOMES:
Participant Body Mass (kg) | Taken at baseline, 6 weeks and 12 weeks/programme completion.
  Participant Body Mass will be measured using calibrated, digital scales.
Participant Body Fat Mass (kg) | Taken at baseline, 6 weeks and 12 weeks/programme completion.
  Participant Body Fat Mass will be measured using the BiodyXpertZMII.
Participant Body Fat Percentage (%) | Taken at baseline, 6 weeks and 12 weeks/programme completion.
  Participant Body Fat Percentage will be measured using the BiodyXpertZMII.
Participant Fat Free Mass (%) | Taken at baseline, 6 weeks and 12 weeks/programme completion.
  Participant Fat Free Mass will be measured using the BiodyXpertZMII.
Participant Body Mass Index (kg/m^2) | Taken at baseline, 6 weeks and 12 weeks/programme completion.
  BMI will be calculated from combining body mass (kg) and participant height (cm).
Participant waist to hip ratio | Taken at baseline, 6 weeks and 12 weeks/programme completion.
  Waist to hip ratio will be calculated from combining measures of waist circumference (cm) and hip circumference (cm).
Participant resting blood pressure (mmHg) | Taken at baseline, 6 weeks and 12 weeks/programme completion.
  Resting diastolic and systolic blood pressure (mmHg) will be taken using a blood pressure monitor.

OTHER OUTCOMES:
Functional Ability (aerobic capacity and endurance) change through Six Minute Walk test | Taken at baseline and 12 weeks/programme completion.
  This will be measured using the Six Minute Walk test and change will be compared within and between participants.
Functional Ability (leg strength and endurance) change through 30s Sit to Stand test | Taken at baseline and 12 weeks/programme completion.
  This will be measured using the 30s Sit to Stand test and change will be compared within and between participants.
Functional Ability (strength) change through hand grip strength test | Taken at baseline and 12 weeks/programme completion.
  This will be measured using the hand grip dynamometer, and change will be compared within and between participants.
Quality of Life and Cost Effectiveness | Taken at baseline, 6 weeks and 12 weeks/programme completion.
  This will be measured using the European Quality of Life Five Dimension Questionnaire (EQ-5D-5L), and change will be compared within and between participants. Scores range from 1-5 with lower scores associated with a better outcome.
Physical Activity | Taken at baseline, 6 weeks and 12 weeks/programme completion.
  This will be measured using the International Physical Activity Questionnaire - Long Form (IPAQ-LF), and change will be compared within and between participants. Scores may be categorised and/or sub scores calculated for each domain where higher scores are associated with better physical activity behaviour.
Exercise Intensity | Three/four times weekly, throughout the 12 week programme, after each exercise session is complete.
  Exercise intensity will be recorded using the Borg Category Ratio (CR-10) scale, and change will be compared to the prescribed programme intensity. Higher scores are associated with a higher exercise intensity.
Exercise Feeling | Three/four times weekly, throughout the 12 week programme, after each exercise session is complete.
  Exercise feeling will be recorded using the Feeling Scale, that ranges from -5 to +5, where -5 indicates feeling 'Very Bad' and +5 indicates feeling 'Very Good'.

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Power, Principal Investigator — Coventry University

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.